CLINICAL TRIAL: NCT02515266
Title: Evaluation of Additional Protein Fortification in Extremely Low Birth Weight Infants Fed Human Milk: PROTSUP Study
Brief Title: Additional Protein Fortification in Extremely Low Birth Weight Infants
Acronym: PROTSUP
Status: Completed | Type: Observational
Sponsor: Hôpital de la Croix-Rousse (Other)
Responsible Party: Principal Investigator, Jean-charles PICAUD, MD, PhD, Head of department of neonatology, Hôpital de la Croix-Rousse
Other Study IDs: 20121
Record Dates: First submitted 2015-07-27; First posted 2015-08-04 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-07

CONDITIONS: Premature Birth; Infant, Extremely Low Birth Weight; Growth Failure
Keywords: protein; growth; head circumference
MeSH Terms: conditions — Premature Birth; Failure to Thrive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: nutrition: protein intake — additional protein fortification of human milk

SUMMARY:
Postnatal growth is a crucial in premature infants as it could be correlated with the long-term cognitive development. Optimal nutritional care is required to reduce the initial weight loss and further growth deficit.

The quantitative objective is to achieve growth that is at least equivalent to that of the fetus (on average 15 g/kg.day (12-18 g/kg.day according to gestational age). Children often grow during difficult 10-15 first days of life, so they accumulate a delay that should compensate them secondarily. Therefore, optimum postnatal growth is rather 20 g/kg.day than 15 g/kg.day.

Individualized fortification of human milk (HM) has been proposed to optimize postnatal growth. Specifically, the lack of protein intake is responsible for sub-optimal postnatal growth in preterm infants.

The objectives of this study are to determine the effectiveness of additional protein fortification (APF) in terms of short-term growth along with the proportion of extremely low birth weight (ELBW) infants requiring APF.

DETAILED DESCRIPTION:
In a retrospective, single-center study, premature infants weighing <1250 g at birth hospitalized in investigators' neonatal intensive care unit in 2012, who were exclusively fed with fortified HM and received APF for >12 consecutive days were included.

Weight gain (g/kg•d) over the previous 7 days was calculated daily based on weight data in patients' electronic medical records. When weight gain was considered insufficient (i.e., below 20 g/kg•d) and the serum urea level was <3 mmol/L, 1 g/kg•d protein was added. Before using the mixture, investigators verified that the osmolality was only slightly increased (from 412 to 422 mOsm/kg).

Growth and digestive tolerance were compared between the week before (Wk0) and 1 and 2 weeks after (Wk1 and Wk2, respectively) the introduction of protein supplement; each participant served as his own control. Change from baseline for body weight was the main outcome. Energy and protein intake during Wk0, Wk1, and Wk2 were calculated. Standard deviation z-scores for growth parameters were calculated 7 days before, at time of protein introduction, and 7 and 14 days after . Changes in Z-scores were calculated. The digestive tolerance score and metabolic tolerance (serum urea) were assessed during Wk0, Wk1, and Wk2 (5).

ELIGIBILITY:
Inclusion Criteria:

* infants weighing <1250 g at birth
* exclusively fed with fortified HM

Exclusion Criteria:

- Severe malformations

Max Age: 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants weighing <1250 g at birth, who were exclusively fed with fortified HM and received additional proteinfortification for >12 consecutive days.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2015-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline body weight z-scores to 1 and 2 weeks after additional protein fortification | One and two weeks after the beginning of additional protein fortification

CONTACTS AND LOCATIONS:
Overall Officials: Jean-charles PICAUD, MD, PhD, Study Director — Hospices Civils de Lyon

REFERENCES:
- [Derived] Picaud JC, Houeto N, Buffin R, Loys CM, Godbert I, Hays S. Additional Protein Fortification Is Necessary in Extremely Low-Birth-Weight Infants Fed Human Milk. J Pediatr Gastroenterol Nutr. 2016 Jul;63(1):103-5. doi: 10.1097/MPG.0000000000001142. PMID 26859094